CLINICAL TRIAL: NCT03921853
Title: Preventing Metabolic Syndrome in Patients With Morbid Obesity by Resistance Training: Reporting Non-responder Prevalence
Brief Title: Resistance Training in Patients With Morbid Obesity
Acronym: ExinMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Los Lagos (Other)
Collaborators: Universidad de La Frontera (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RP08042019
Record Dates: First submitted 2019-04-08; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Morbid Obesity; Obesity; Physical Activity; Metabolic Syndrome; Risk Factor, Cardiovascular
MeSH Terms: conditions — Obesity, Morbid; Obesity; Motor Activity; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: We will compare a control group with obesity with another experimental group with morbid obesity in the metabolic syndrome parameters.
Who Masked: Investigator
Masking Description: According with the availability and the feasibility of the enrolment's requirements, patients will be allocated to a control group with obesity, and another with morbid obesity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active comparator (Active Comparator): Control group with obesity under Resistant Training
  Interventions: Other: Behavioral
- Experimental group with morbid obesity (Experimental): Experimental group with morbid obesity under Resistant Training
  Interventions: Other: Behavioral

INTERVENTIONS:
Other: Behavioral — The 20-week RT program will consist of three sessions per week, each lasting for 1 hour that will be applied to both control obese (CG) and morbid obese (MO) group. All sessions will start with 15 minutes warm-up with continuous walking and joint mobility and flexibility exercises, 5 minutes of cool down and stretching, in order for preventing injuries. Sessions will include 4 to 8 RT exercises targeting different muscle groups; 1. forearm, 2. knee flexors and 3. extensors, 3. trunk, 4. chest, 5. shoulder elevators, 6. horizontal shoulder flexors and 7. extensors, and 8. plantar flexors. The exercises for each muscle group will be performed in 3 sets of as many repetitions (continuous concentric/eccentric voluntary contraction) possible in 1 minute followed by 2.0 minutes of passive recovery. Before the RT program, each participant will be measure using the subjective modified Borg scale (1-10 points), in order of identifying the muscle failure into 1 minute of exercise.
  Other Names: Resistant training intervention

SUMMARY:
The researchers will conduct a study for avoiding the metabolic syndrome in morbid obese patients. Thus, the aim of the present will be determine the effects of a resistance training programme (RT) in preventing or attenuating metabolic syndrome (MetS) in patients with morbid obesity. A second aim will be report the prevalence of non-responders in terms of improvements in MetS markers and other co-variables considered.

DETAILED DESCRIPTION:
The prevalence of metabolic syndrome (MetS) and cardiovascular disease is expected to rise along with the global obesity epidemic. MetS is a cluster of clinical risk factors, including abdominal (visceral) obesity, hypertension, elevated serum triglycerides, low serum high-density lipoprotein (HDL) and hyperglycaemia.The MetS for example, significantly decreases the life expectancy of individuals with morbid obesity and increases the disease burden and economic costs associated with healthcare. In this sense, more recently, there was reported that body mass index (BMI) and fat distribution showed higher associations with inflammation, fat indices, and more prevalence of MetS in morbidly obese subjects, claiming for an early prevention of the MetS in the morbid obese state.

Exercise training has proven to be effective in inducing a clinically significant weight loss and reducing cardiovascular risk. Exercise have reported to be associated with increased muscle mass, decreased body fat, and improved metabolic profile (i.e., improved glucose control and lipid levels). In addition, supervised RT improved muscle strength and functional capacity in patients with obesity undergoing bariatric surgery. However, although RT has been widely studied in obesity, there is little information in the morbid obesity. On the other hand, there is poor knowledge similarly, about the interindividual variability to exercise training in terms of responders and non-responders (NR). Thus, considering the poor knowledge about the MetS prevention in morbid obese patients, as well as the little information about Responders and Non-Responders for improving MetS outcomes, the aim of this study will be determine the effects of a RT program on cardio-metabolic outcomes of MetS in patients with morbid obesity. A second aim will be report the prevalence of non-responders in terms of the effects of resistance training on MetS markers and other health-related variables.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Older than 18 and younger and ≤65 years of age.
* With risk factors to Metabolic syndrome
* With obesity and morbid obesity condition
* Medical authorization by a physician.

Exclusion Criteria:

* Physical limitations (e.g., restricting injuries of the musculoskeletal system, or dependent of a third person).
* Exercise-related dyspnoea or respiratory alterations.
* Chronic heart disease with any worsening in the last month.
* Adherence rate of less than 80% of the total interventions.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | Change from Baseline Fasting glucose at 20-weeks of Resistant Training
  Component of the Metabolic Syndrome
High density lipoprotein | Change from Baseline High density lipoprotein at 20-weeks of Resistant Training
  Component of the Metabolic Syndrome
Systolic blood pressure and diastolic blood pressure | from Baseline Systolic blood pressure and diastolic blood after 20-weeks of Resistant Training
  Component of the Metabolic Syndrome
Waist circumference | Change from Baseline Waist circumference at 20-weeks of Resistant Training
  Component of the Metabolic Syndrome
Triglycerides | Change from Baseline Triglycerides at 20-weeks of Resistant Training
  Component of the Metabolic Syndrome

SECONDARY OUTCOMES:
Body mass index | Change from Baseline Body mass index at 20-weeks of Resistant Training
  Anthropometric
Body mass | Change from Baseline Body mass at 20-weeks of Resistant Training
  Anthropometric
Total cholesterol | Change from Baseline Total cholesterol at 20-weeks of Resistant Training
  Measured by plasma sample
Low density lipoprotein | Change from Baseline Low density lipoprotein at 20-weeks of Resistant Training
  Measured by plasma sample
Six minutes walking test | Change from Baseline Six minutes walking test density lipoprotein at 20-weeks of Resistant Training
  Endurance performance
One maximum repetition of biceps curl | Change from Baseline One maximum repetition of biceps curl at 20-weeks of Resistant Training
  Strength Performance
Handgrip muscle strength | Change from Baseline Handgrip muscle strength at 20-weeks of Resistant Training
  Muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Cristian ALvarez, PhD, Study Director — Universidad de Los Lagos
Locations (1):
- Cristian ALvarez, Osorno, Llanquihue, Chile

IPD SHARING:
Plan to Share IPD: No
The participants information will be available by e-mail according with researchers requirements.

REFERENCES:
- [Derived] Delgado-Floody P, Alvarez C, Lusa Cadore E, Flores-Opazo M, Caamano-Navarrete F, Izquierdo M. Preventing metabolic syndrome in morbid obesity with resistance training: Reporting interindividual variability. Nutr Metab Cardiovasc Dis. 2019 Dec;29(12):1368-1381. doi: 10.1016/j.numecd.2019.07.002. Epub 2019 Jul 12. PMID 31383503

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT03921853/Prot_SAP_000.pdf